CLINICAL TRIAL: NCT06656143
Title: Effects of Diaphragmatic Myofascial Release on Chest Expansion and Heart Rate in Patients With Thoracic Kyphosis
Brief Title: Diaphragmatic Myofascial Release Techinque on Chest Expansion and Heart Rate in Patients Having Thoracic Kyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/014375 Ayeza Naser
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Thoracic Kyphosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Myofascial release (Experimental): Myofascial release of the diaphragm is an intervention intended to indirectly stretch the diaphragm muscle fibers to reduce muscle tension, normalize fiber length, and promote the efficiency of muscle contraction.
  Interventions: Other: Diaphragmatic Myofascial Release
- Traditional Physical therapy (Active Comparator): Strengthening Deep Cervical Flexors Strengthening Shoulder Retractors Stretch Cervical Extensors Stretch Pectoralis Muscle
  Interventions: Other: Traditional Physical therapy

INTERVENTIONS:
Other: Traditional Physical therapy — The exercise program included the strengthening of the deep cervical flexor and shoulder retractor muscles and also stretching of the pectoralis and cervical extensor muscles.
  (3 sets of 12 repetitions) Strengthening Deep Cervical Flexors Lying chin tuck Lying chin tuck with head lift. Strengthening Shoulder Retractors Standing shoulder pull back with elastic Shoulder pull back with weight Stretch Cervical Extensors Chin drop Stretch Pectoralis Muscle Bilateral Pectoral stretch
  Arms: Traditional Physical therapy
Other: Diaphragmatic Myofascial Release — To release the diaphragm, the patient was positioned in the supine position. The therapist stood at the head of the patient. The therapist made manual contact bilaterally under the costal cartilages of the lower ribs (7th to 10th) with hypothenar regions of the hands and last three fingers. During the patient's inspiration, the therapist was gently pulling the points of hands contacts toward the head and slightly laterally, while elevating the ribs simultaneously. During exhalation, the therapist deepened hand contacts towards the inner costal margins Exercise Program (3 sets of 12 reps) Strengthening deep cervical flexors Strengthening shoulder retractors Stretching Cervical Extensors Stretching Pectoralis Muscle
  Arms: Diaphragmatic Myofascial release

SUMMARY:
The air of this RCT is to evaluate the effects Diaphragmatic Myofascial Release technique on chest expansion and heart rate in patients with thoracic kyphosis

DETAILED DESCRIPTION:
This study focus on diaphragmatic release technique along with conventional therapy is more effective in improving chest expansion and with im-proved chest expansion, heart rate and blood pressure is also improved because tho-racic kyphosis impacts the way of heart and lung function creating stress response and increasing heart rate and blood pressure. Lung capacity is also reduced in indi-viduals with thoracic kyphosis. Postural alterations of thoracic spine result in im-paired chest expansion and length tension curve of diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Both male and females
* age 18-40 years
* patients who consented to the purposes of this study and participated voluntarily.
* patients with thoracic kyphosis ≥40

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.
* Vertebrobasilar insufficiency, rib fracture, rib dislocation and/or signs of serious pathology (e.g., malignancy, inflammatory disorder, infection);
* History of cervical spine surgery in previous 12 months
* Signs of cervical radiculopathy or myelopathy; and vascular syndromes such as basilar insufficiency.
* Patients with diagnosed any respiratory condition.
* Patient diagnosed with hypertension or taking any medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Chest Expansion | 3rd week
  Diaphragm is facially and mechanically attached to thoracic spine, so releasing tension in diaphragmatic muscles will improve biomechanics, resulting in greater chest expansion and improving heart rate.
Heart Rate | 3rd week
  Diaphragm a thin, flat muscle that separates the thoracic and abdominal cavity, is the primary muscle of respiration, which plays significant role in breathing and physiological regulation. Hyper kyphosis negatively affects chest expansion and heartrate by causing limited mobility in thoracic cage. Diaphragm is facially and mechanically attached to thoracic spine, so releasing tension in diaphragmatic muscles will improve biomechanics, resulting in greater chest expansion and improving heart rate

SECONDARY OUTCOMES:
Thoracic Kyphosis | 3rd week
  Kyphosis is an abnormal convex curvature in thoracic spine, certain factors such as neuromuscular disorders, congenital anomalies and positional difficulties trigger development of kyphotic posture. Thoracic kyphosis affects the physiological and anatomical feature of the human body

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila Yaqub, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singla D, Veqar Z. Association Between Forward Head, Rounded Shoulders, and Increased Thoracic Kyphosis: A Review of the Literature. J Chiropr Med. 2017 Sep;16(3):220-229. doi: 10.1016/j.jcm.2017.03.004. Epub 2017 Sep 28. PMID 29097952
- [Background] Park SJ, Kim SH, Kim SH. Effects of Thoracic Mobilization and Extension Exercise on Thoracic Alignment and Shoulder Function in Patients with Subacromial Impingement Syndrome: A Randomized Controlled Pilot Study. Healthcare (Basel). 2020 Sep 2;8(3):316. doi: 10.3390/healthcare8030316. PMID 32887287
- [Background] Lewis JS, Valentine RE. Clinical measurement of the thoracic kyphosis. A study of the intra-rater reliability in subjects with and without shoulder pain. BMC Musculoskelet Disord. 2010 Mar 1;11:39. doi: 10.1186/1471-2474-11-39. PMID 20193055